CLINICAL TRIAL: NCT03476486
Title: A Pilot Study to Evaluate the Effectiveness of Ultrasound Guided Looped Thread Carpal Tunnel Release
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00060817
Record Dates: First submitted 2018-03-17; First posted 2018-03-26 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2018-03

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Intervention Model Description: controlled interventional clinical trial
Who Masked: Outcomes Assessor
Masking Description: single blind masking (assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): The hand that was subject to thread carpal tunnel release surgery
  Interventions: Procedure: Thread carpal tunnel release
- Control (No Intervention): The hand that was not treated

INTERVENTIONS:
Procedure: Thread carpal tunnel release — Ultrasound-guided percutaneous minimally invasive thread carpal tunnel release using a looped thread technique
  Arms: Treatment

SUMMARY:
Carpal tunnel syndrome occurs when a nerve gets pinched as it passes through a confined tunnel within the wrist and hand. It is the most commonly pinched nerve and often results in disabling hand numbness, tingling, pain and weakness. For moderate and severe cases, an operation is often performed that cuts the ligament that presses on the nerve. This surgery is generally very successful but involves a 2-5 cm long incision at the base of the palm. Recovery from the surgery usually takes 3-8 weeks. Ultrasound provides a clear noninvasive way of looking at the contents of the carpal tunnel. A technique has been developed whereby a wire thread is looped around the ligament using a needle guided by ultrasound. The ligament is cut by the wire below the surface of the skin. This technique results in 2 needle puncture holes instead of the open incision of the traditional surgery. The investigators have completed research on this technique in cadavers. It was confirmed that complete or almost complete cutting of the ligament can be safely and predictably accomplished. This research will look at the effectiveness of this looped thread technique of carpal tunnel release on patients who have carpal tunnel syndrome. Specifically, participants will be required to: 1. rate the severity of their carpal tunnel syndrome symptoms and disability using a standard questionnaire, 2. measure hand sensation, 3. measure pinch and grip strength tests of their hands, 4. undergo ultrasound measurements of the size of the pinched nerve at the carpal tunnel, and 5. undergo electrical tests to measure the nerves ability to conduct impulses across the carpal tunnel. These will be measured before the looped wire procedure and at 3 and 6 months following the procedure. Recovery time will also be measured.

DETAILED DESCRIPTION:
Objectives: to evaluate the effectiveness and safety of a minimally invasive ultrasound-guided looped thread technique of carpal tunnel release

Background: Carpal tunnel syndrome (CTS) is the most common peripheral entrapment neuropathy, having a prevalence of 3.7%. CTS is the 2nd leading worktime loss condition. Open surgical decompression of the carpal tunnel is an evidence-based and commonly performed treatment for moderate to severe cases, predictably providing long-term symptom relief. This surgical technique involves placing a 2-5 cm long longitudinal incision at the palm, incising the skin, subcutaneous tissue, palmar fascia, palmaris longus tendon (if present) and transverse carpal ligament under direct visualization. After 3-8 weeks of recovery, most patients experience excellent relief of symptoms and improvement in hand function. On occasion, the procedure is complicated by nerve damage, scar or pillar pain. A variety of strategies have been devised to minimize the invasive nature of carpal tunnel release in hopes to reduce post procedure pain, weakness and recovery time. In the late 1980s, an endoscopic release technique was devised. A recent meta-analysis of existing randomized control trials comparing open to endoscopic release found endoscopic release to provide better early recovery of grip and pinch strength, less scar tenderness and earlier returned to work (~9 days). There was a similar risk of pillar pain and reoperation, and a higher risk of nerve injury (mostly transient neurapraxia). The development of high-resolution ultrasound scanning allows detailed visualization of the carpal tunnel and its contents. Hydrodissection, the injection of fluid during ultrasound visualization, adds to image clarity of both the contents of the carpal tunnel as well as the location of operative instruments. A few minimally invasive ultrasound-guided percutaneous carpal tunnel release techniques have been described. The cutting instruments have included needle tip, knife, saws blades, and thread. Initial results of these techniques suggest that they are feasible, safe, effective and are associated with short recovery times. The most recently described minimally invasive technique involves percutaneously looping a cutting thread around the transverse carpal ligament using a needle under ultrasound guidance. By reciprocally sliding the 2 ends of the thread back and forth like a Gigli saw, the transverse carpal ligament is transected. Only 2 needle puncture site are required. The looped thread carpal tunnel release (TCTR) procedure was initially performed on a single cadaveric hand and dissection demonstrated complete transection of the transverse carpal ligament and no injury to other structures. The authors then performed the same procedure on 34 hands of 20 patients. The primary outcome measure was the Levine-Katz questionnaire completed 3 months postprocedure. The questionnaire scores were compared to those reported in the literature for open and endoscopic release techniques and were found to be similar. No post TCTR complications were reported. Our research group has recently completed a cadaveric evaluation of this technique and found that ultrasound accurately defines the critical boundries and contents of the carpal tunnel in all cases, complete or near-complete transection of the transverse carpal ligament was achieved and no trauma was sustained by any structure within the carpal tunnel other than the transverse carpal ligament.

Procedure/Methods: subjects with clinical and electrophysiologically confirmed CTS from the practice of the principal investigator will be invited to participate. The 1st phase of this study will involve TCTR of 5 carpal tunnels. Within a month prior to and at 3 and 6 months post procedure the following outcome measures will be collected: subjective measure of symptom and functional limitation severity (Boston Carpal Tunnel Questionnaire); monofilament hand sensibility testing, grip and pinch strength; median nerve cross-sectional area measurement at the carpal tunnel inlet using ultrasound; and electrophysiologic function of the median nerve across the carpal tunnel (motor and sensory conduction velocities and amplitudes). At weekly intervals for the 1st month, each subject will also be contacted to report on their recovery (return to everyday activities including work) and any adverse effects/complications. The Boston Carpal Tunnel Questionnaire will also be completed at 1 month post TCTR. Assuming no serious complications are encountered from the initial 5 procedures, and upon approval from the supervising Data and Safety Monitoring Board, 15 additional carpal tunnels will undergo TCTR and the same outcome measures will be recorded. The outcome data will be analyzed using a repeated measures Analysis of Variance (Boston Carpal Tunnel Questionnaire; monofilament hand sensibility;grip and pinch strength; median nerve cross-sectional area; median nerve motor and sensory conduction velocities and amplitudes) and descriptive statistics (recovery duration and adverse effects/complications).

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* symptoms (hand numbness, tingling, weakness or pain; symptom aggravation with repetitive or sustained gripping; nocturnal symptom exacerbation) and signs (hand sensory disturbance or weakness; positive median nerve Tinel's sign or Phalen's test) compatible with carpal tunnel syndrome
* symptom duration >3 months refractory to conservative treatment (i.e. wrist splints, activity modification, NSAID, +/- intracarpal tunnel corticosteroid injection)
* nerve conduction study abnormalities compatible with moderate to severe median neuropathy at the carpal tunnel (motor and sensory conduction slowing across the carpal tunnel +/- evidence of axonal loss)
* signed informed consent

Exclusion Criteria:

* ultrasound identifies a bifid median nerve or persistent median artery at the carpal tunnel inlet
* Clinical or electrophysiologic evidence of a neurologic disorder of the upper extremity besides carpal tunnel syndrome (i.e. proximal median neuropathy; ulnar or radial neuropathy, brachial plexopathy, cervical radiculopathy or generalized polyneuropathy)
* Inability to understand the informed consent or the Boston Carpal Tunnel Questionnaire
* Coagulopathy or anticoagulation that cannot be stopped for the carpal tunnel release procedure
* Local anesthetic allergy
* systemic infection or a local infection at the procedure site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-05-20 (Actual); Primary Completion 2018-01-20 (Actual); Study Completion 2018-01-20 (Actual)

PRIMARY OUTCOMES:
Early recovery | 1st month following the thread carpal tunnel release surgery
  At weekly intervals for the 1st month ,each subject will also be contacted to report on their recovery (return to everyday activities including work) and any adverse effects/complications
Boston Carpal Tunnel Questionnaire | a month prior to and at 3 and 6 months post procedure
  subjective measure of symptom and functional limitation severity. Symptom and function subscale scores were summed (score range 2-10 with 2=asymptomatic and 10=severely symptomatic).
Hand sensation | a month prior to and at 3 and 6 months post procedure
  monofilament hand sensibility testing
grip and pinch strength | a month prior to and at 3 and 6 months post procedure
  Grip strength measured using a hand grip dynamometer; pinch strength measured with a pinch dynamometer
Median nerve cross-sectional area | a month prior to and at 3 and 6 months post procedure
  median nerve cross-sectional area measurement at the carpal tunnel inlet using ultrasound
Median nerve electrophysiologic function | a month prior to and at 3 and 6 months post procedure
  electrophysiologic function of the median nerve across the carpal tunnel (motor and sensory conduction velocities and amplitudes).
Subject satisfaction | 3 and 6 months post thread carpal tunnel release
  Global satisfaction score

CONTACTS AND LOCATIONS:
Overall Officials: Robert Burnham, Principal Investigator — University of Alberta

IPD SHARING:
Plan to Share IPD: No